CLINICAL TRIAL: NCT02497391
Title: A Bioequivalence Study in Healthy Subjects Administered Evacetrapib Tablets of Varying Particle Sizes
Brief Title: A Study of Different Particle Sizes of Evacetrapib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14629; I1V-MC-EIBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Results first posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Healthy
MeSH Terms: interventions — evacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Evacetrapib Reference (R) (Experimental): Single oral dose of 130 mg evacetrapib tablet given one time during one study period.
  Interventions: Drug: Evacetrapib
- Evacetrapib Test 1 (T1) (Experimental): Single oral dose of 130 mg evacetrapib tablet given one time during one study period.
  Interventions: Drug: Evacetrapib
- Evacetrapib Test 2 (T2) (Experimental): Single oral dose of 130 mg evacetrapib tablet given one time during one study period.
  Interventions: Drug: Evacetrapib

INTERVENTIONS:
Drug: Evacetrapib — administered orally
  Other Names: LY2484595

SUMMARY:
The purpose of this study is to determine if there is any difference in the way the body handles 3 types of evacetrapib tablets with different particle sizes. Information about any side effects will also be collected. This study will consist of 3 study periods. Participants will be dosed 3 times during the entire study. Each study period will consist of an inpatient stay for 3 days - the day before dosing (Day -1), dosing day (Day 1) and the day after dosing (Day 2). Then participants will be asked to return to the clinical research unit (CRU) daily for outpatient appointments up to Day 8. The overall length of this study is about 7 weeks from first dose to end of study. Screening will take place within 28 days prior to the first dose of evacetrapib and follow-up will take place 21 days after the last dose of evacetrapib.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy participants of non-child bearing potential
* Have a body mass index of 18 to 32 kilograms per square meter (kg/m^2)
* Must be willing to make oneself available for the whole study and be willing to follow study procedures

Exclusion Criteria:

* Have known allergies to evacetrapib, compounds or components related to this drug, or have a history of significant allergic reactions of another origin.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 6 treatment sequences in a crossover design with 3 treatments; reference, test 1 and test 2. There was a washout period of ≥14 days between each dose. Participants were dosed 3 times during the entire study in periods 1, 2 and 3.
Groups:
- Sequence 1 (R/T1/T2): Single oral dose of evacetrapib 130 mg tablet given one time during one study period as a evacetrapib reference (R1), evacetrapib test 1 (T1) or evacetrapib test 2 (T2) formulation.
  All participants received one tablet in Period 1: R Period 2: T1 Period 3: T2
- Sequence 2 (T1/T2/R): Single oral dose of evacetrapib 130 mg tablet given one time during one study period as a evacetrapib reference (R1), evacetrapib test 1(T1) or evacetrapib test 2 (T2) formulation.
  All participants received one tablet in Period 1: T1 Period 2: T2 Period 3: R
- Sequence 3 (T2/R/T1): Single oral dose of evacetrapib 130 mg tablet given one time during one study period as a evacetrapib reference (R1), evacetrapib test 1 (T1) or evacetrapib test 2 (T2) formulation.
  All participants received one tablet in Period 1: T2 Period 2: R Period 3: T1
- Sequence 4 (T2/T1/R): Single oral dose of evacetrapib 130 mg tablet given one time during one study period as a evacetrapib reference (R1), evacetrapib test 1 (T1) or evacetrapib test 2 (T2) formulation.
  All participants received one tablet in Period 1: T2 Period 2: T1 Period 3: R
- Sequence 5 (R/T2/T1): Single oral dose of evacetrapib 130 mg tablet given one time during one study period as a evacetrapib reference (R1), evacetrapib test 1 (T1) or evacetrapib test 2 (T2) formulation.
  All participants received one tablet in Period 1: R Period 2: T2 Period 3: T1
- Sequence 6 (T1/R/T2): Single oral dose of evacetrapib 130 mg tablet given one time during one study period as a evacetrapib reference (R1), evacetrapib test 1 (T1) or evacetrapib test 2 (T2) formulation.
  All participants received one tablet in Period 1: T1 Period 2: R Period 3: T2
Period: Period 1 (14 Days)
Arm/Group | Sequence 1 (R/T1/T2) | Sequence 2 (T1/T2/R) | Sequence 3 (T2/R/T1) | Sequence 4 (T2/T1/R) | Sequence 5 (R/T2/T1) | Sequence 6 (T1/R/T2)
Started | 16 | 15 | 16 | 16 | 16 | 16
Received at Least 1 Dose of Study Drug | 16 | 15 | 16 | 16 | 16 | 16
Completed | 16 | 15 | 16 | 16 | 16 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (14 Days)
Arm/Group | Sequence 1 (R/T1/T2) | Sequence 2 (T1/T2/R) | Sequence 3 (T2/R/T1) | Sequence 4 (T2/T1/R) | Sequence 5 (R/T2/T1) | Sequence 6 (T1/R/T2)
Started | 16 | 15 | 16 | 16 | 16 | 16
Completed | 12 | 14 | 13 | 13 | 14 | 13
Not Completed | 4 | 1 | 3 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 3 | 1 | 2 | 3 | 2 | 3
Period: Period 3 (14 Days)
Arm/Group | Sequence 1 (R/T1/T2) | Sequence 2 (T1/T2/R) | Sequence 3 (T2/R/T1) | Sequence 4 (T2/T1/R) | Sequence 5 (R/T2/T1) | Sequence 6 (T1/R/T2)
Started | 12 | 14 | 13 | 13 | 14 | 13
Completed | 12 | 13 | 12 | 13 | 13 | 13
Not Completed | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Participants received a single dose of 130 mg evacetrapib tablet (a total of 3 doses of evacetrapib) given one time during each study period.
Arm/Group | Overall Participants
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 92
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 95

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Evacetrapib
Time Frame: Predose on Day 1,and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 Hours Postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nangram/milliliter (ng/mL)
Groups:
- Evacetrapib Reference (R); Evacetrapib Test 1 (T1); Evacetrapib Test 2 (T2): Single oral dose of evacetrapib 130 mg tablet given one time during one study period.
Arm/Group | Evacetrapib Reference (R) | Evacetrapib Test 1 (T1) | Evacetrapib Test 2 (T2)
Number analyzed (Participants) | 84 | 81 | 85
nangram/milliliter (ng/mL) | 983 (78) | 1170 (56) | 1120 (66)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Evacetrapib
Time Frame: Predose on Day 1,and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 Hours Postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram·hour/milliter (ng·h/mL)
Arm/Group | Evacetrapib Reference (R) | Evacetrapib Test 1 (T1) | Evacetrapib Test 2 (T2)
Number analyzed (Participants) | 84 | 81 | 85
nanogram·hour/milliter (ng·h/mL) | 14700 (53) | 16100 (45) | 15500 (49)

ADVERSE EVENTS:
Arm/Group | Evacetrapib Reference (R) | Evacetrapib Test 1 (T1) | Evacetrapib Test 2 (T2)
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/81 | 0/85
Other Adverse Events (participants affected / at risk) | 33/84 | 22/81 | 23/85
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib Reference (R) (N=84) | Evacetrapib Test 1 (T1) (N=81) | Evacetrapib Test 2 (T2) (N=85)
Catheter site related reaction (General disorders) | 13 (13) | 9 (9) | 2 (2)
Vessel puncture site bruise (General disorders) | 16 (17) | 12 (13) | 20 (21)
Headache (Nervous system disorders) | 6 (6) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days